CLINICAL TRIAL: NCT07211815
Title: Dosimetric Differences and Clinical Significance Analysis Between Body Gamma Knife and VMAT Radiotherapy for Primary Liver Cance
Status: Not yet recruiting | Type: Observational
Sponsor: Chifeng Tumor Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CFSZLYY - FLK - 2025 - 001
Record Dates: First submitted 2025-09-22; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Primary Liver Cancers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gamma Knife Treatment Group: Patients in this group receive body gamma knife radiotherapy. The treatment utilizes fixed radiation sources, and the treatment couch moves to each treatment target. A 50% isodose curve covers at least 95% of the Planning Target Volume (PTV), and this modality is applied for radiotherapy of locally advanced primary liver cancer.
- Accelerator Treatment Group: Patients in this group receive radiotherapy with an accelerator (applying VMAT technology). Based on the tumor's location and surrounding organs at risk, beam angles and the number of fields are selected. The prescription dose curve covers 95% of the Planning Target Volume (PTV), and this method is used for radiotherapy of locally advanced primary liver cancer.

SUMMARY:
To fill in the "Brief Summary" field, you need to provide clear, easy-to-understand information about the study for patients, families, and healthcare providers. Here's a suggested summary:

This study compares the dosimetric features and clinical effects of body gamma knife and VMAT radiotherapy for locally advanced primary liver cancer. We retrospectively analyze 20 patients from Chifeng Tumor Hospital who cannot or refuse surgery. For each patient, we will develop both body gamma knife and VMAT radiotherapy plans. Then, we'll compare the dose distribution in the tumor target (including conformity index and homogeneity index) and the radiation exposure to organs at risk (such as the spinal cord, stomach, and liver). The goal is to find out which radiotherapy approach is more beneficial, so patients, families, and healthcare teams can better understand how this research supports treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years.
* Clinically or pathologically confirmed primary liver cancer; unsuitable for or - refusing surgery, with single tumor diameter ≤5 cm and ≤5 nodules.
* ECOG PS score 0-1.
* Liver function: Child-Pugh grade A or B.
* Prothrombin time (PT) < 4 seconds above the normal control range.
* No hepatic encephalopathy or moderate to large ascites.
* Renal and cardiopulmonary function basically normal.
* Gastroscopy findings: no severe esophageal varices or active peptic ulcer.
* Hemoglobin ≥90 g/L, WBC ≥3.0×10⁹/L, neutrophil ≥1.5×10⁹/L, platelet ≥40×10⁹/L.
* No obvious cachexia; life expectancy > 3 months.
* Not pregnant; no HIV or syphilis infection.
* Able to understand the study and sign informed consent.

Exclusion Criteria:

* History of portal hypertension, esophageal variceal bleeding, or related conditions.
* History of anti-RHCC treatment or spontaneous tumor rupture.
* Postoperative pathology indicates metastatic cancer or other primary cancers.
* Cerebrovascular accident within 6 months before enrollment.
* Severe lung disease; serum creatinine > 1.25×the upper normal limit.
* Poorly controlled acute or active infection; severe mental illness.
* Suspected systemic or local lymphadenopathy on imaging.
* Pregnant or lactating women; presence of other serious underlying diseases.
* Currently participating in other clinical trials; refusal to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced primary liver cancer (unsuitable for/refusing surgery, meeting inclusion & not exclusion criteria), aged 18-75 years, from Chifeng Tumor Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Conformity Index Comparison: Body Gamma Knife vs. VMAT for Locally Advanced Primary Liver Cancer | Within 1 month after completion of radiotherapy planning
  Compare the conformity index (a dosimetric measure of how well radiation conforms to the target volume) between body gamma knife and VMAT radiotherapy in patients with locally advanced primary liver cancer.

SECONDARY OUTCOMES:
Gradient Index Comparison: Body Gamma Knife vs. VMAT for Locally Advanced Primary Liver Cancer | Within 1 month after completion of radiotherapy planning
  Compare the gradient index (a dosimetric measure of dose fall-off outside the target volume) between body gamma knife and VMAT radiotherapy in patients with locally advanced primary liver cancer.
Homogeneity Index Comparison: Body Gamma Knife vs. VMAT for Locally Advanced Primary Liver Cancer | Within 1 month after completion of radiotherapy planning
  Compare the homogeneity index (a dosimetric measure of dose uniformity within the target volume) between body gamma knife and VMAT radiotherapy in patients with locally advanced primary liver cancer.
Liver V20 Comparison: Body Gamma Knife vs. VMAT for Locally Advanced Primary Liver Cancer | Within 1 month after completion of radiotherapy planning
  Compare the volume of liver receiving 20 Gy (V20) between body gamma knife and VMAT radiotherapy in patients with locally advanced primary liver cancer.
Liver Mean Dose (Dmean) Comparison: Body Gamma Knife vs. VMAT for Locally Advanced Primary Liver Cancer | Within 1 month after completion of radiotherapy planning
  Compare the mean dose (Dmean) to the liver between body gamma knife and VMAT radiotherapy in patients with locally advanced primary liver cancer.
Liver V5 Comparison: Body Gamma Knife vs. VMAT for Locally Advanced Primary Liver Cancer | Within 1 month after completion of radiotherapy planning
  Compare the volume of liver receiving 5 Gy (V5) between body gamma knife and VMAT radiotherapy in patients with locally advanced primary liver cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Chifeng Tumor Hospital, Chifeng, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol